CLINICAL TRIAL: NCT04273178
Title: Feasibility and Outcome of Anti-fungal Prophylaxis With an Escalation Pattern for Patients Undergoing Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Escalation Antifungal Prophylaxis for Patients Undergoing Allogeneic Hematopoietic Stem Cell Transplantation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Jiong HU, Head of Blood and Marrow Transplantation Program, Principle Investigator, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2019-BMT-Prophyfungal
Record Dates: First submitted 2020-02-14; First posted 2020-02-17 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2021-11

CONDITIONS: Fungal Infection
Keywords: fungal infection, stem cell transplantation, prophylaxis
MeSH Terms: conditions — Mycoses

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Escalating prophylaxis (Experimental): For all patients without documented proven or probable invasive fungal disease (IFD), patients will receive fluconazole during the treatment in the laminar air flow units (LAF). After discharged from LAF units, patients will receive anti-mold prophylaxis in case of haplo-identical or HLA-matched unrelated donor transplantation to d+100 without active acute GVHD (aGVHD). In case of active aGVHD, the prophylaxis treatment will be extended until recovery of aGVHD and tapering of immunosuppression. In case of HLA-matched sibling donor, fluconazole will be continued to d+100 and anti-mold prophylaxis will be given in case of active aGVHD.
  Interventions: Drug: Escalating prophylaxis

INTERVENTIONS:
Drug: Escalating prophylaxis — For all patients without documented proven or probable invasive fungal disease (IFD), patients will receive fluconazole during the treatment in the laminar air flow units (LAF). After discharged from LAF units, patients will receive anti-mold prophylaxis in case of haplo-identical or HLA-matched unrelated donor transplantation to d+100 without active acute GVHD (aGVHD). In case of active aGVHD, the prophylaxis treatment will be extended until recovery of aGVHD and tapering of immunosuppression. In case of HLA-matched sibling donor, fluconazole will be continued to d+100 and anti-mold prophylaxis will be given in case of active aGVHD.

SUMMARY:
This is single arm study to evaluate an escalation anti-fungal prophylaxis protocol for patients undergoing allogeneic stem cell transplantation. For all patients without documented proven or probable invasive fungal disease (IFD), patients will receive fluconazole during the treatment in the laminar air flow units (LAF). After discharged from LAF units, patients will receive anti-mold prophylaxis in case of haplo-identical or HLA-matched unrelated donor transplantation to d+100 without active acute GVHD (aGVHD). In case of active aGVHD, the prophylaxis treatment will be extended until recovery of aGVHD and tapering of immunosuppression. In case of HLA-matched sibling donor, fluconazole will be continued to d+100 and anti-mold prophylaxis will be given in case of active aGVHD.

DETAILED DESCRIPTION:
Based on CAESAR study, the IFD incidence increased significantly in patients with unrelated donor or hallo-donor HSCT after patients being discharged from LAF units. The overall incidence of IFD in patients with HLA-matched sibling donor remain low unless in patients with active aGVHD. In this single-arm prospective study, we plan to evaluate the feasibility and effect of an escalation anti-fungal prophylaxis protocol for patients undergoing allogeneic stem cell transplantation. For all patients without documented proven or probable invasive fungal disease (IFD), patients will receive fluconazole during the treatment in the laminar air flow units (LAF). After discharged from LAF units, patients will receive anti-mold prophylaxis in case of haplo-identical or HLA-matched unrelated donor transplantation to d+100 without active acute GVHD (aGVHD). In case of active aGVHD, the prophylaxis treatment will be extended until recovery of aGVHD and tapering of immunosuppression. In case of HLA-matched sibling donor, fluconazole will be continued to d+100 and anti-mold prophylaxis will be given in case of active aGVHD.

ELIGIBILITY:
Inclusion Criteria:

* patients undergo allogeneic HSCT
* Conditioning regimens: myelo-ablative, reduced toxicity
* No proven or probable IFD before HSCT
* No allergy to fluconazole, voriconazle and posaconazole
* Inform consent given

Exclusion Criteria:

* Imparied liver function with (AST or ALT>3ULN, TBil >2ULN)

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 175 (Estimated)
Dates: Start 2020-01-15 (Actual); Primary Completion 2022-01-15 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of IFD | day 180 after transplantation
  Proven and probable diagnosis of IFD

SECONDARY OUTCOMES:
Incidence of IFD2 | day 180 after transplantation
  Proven, probable and possible IFD
Incidence of IFD associated mortality | day 180 after transplantation
  Documentation of death due to proven, probable and possible IFD
Incidence of nor-relapse mortality (NRM) | day 180 after transplantation
  Documentation of death not due to disease relapse or progression

CONTACTS AND LOCATIONS:
Overall Officials: Jiong Hu, Principal Investigator — Ruijin Hospital
Locations (1):
- Blood & Marrow Transplantation Center, RuiJin Hospital, Shanghai, Shanghai Municipality, China